CLINICAL TRIAL: NCT06528925
Title: Effect of Virtual Reality Goggles on Pain, Anxiety and Hemodynamic Variables During Urodynamics: A Randomized Controlled Study
Brief Title: Effect of Virtual Reality Goggles on Pain, Anxiety and Hemodynamic Variables During Urodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Dr. Research Assistant, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TU-BOZKUL-008
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Virtual Goggles; Urodynamics; Pain; Anxiety; Hemodynamic Variables
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-arm (1:1), randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The information showing that the patients included in the research sample are assigned to group A and B according to the randomization table will be placed in an opaque envelope. This envelope will be kept by the researcher (GAU) and when the researchers (GB and EKD) go to the patient for the application, they will open the envelope after filling out the "Informed Consent Form" and learn which group the patient is in. While the researchers (GB and EKD) will be blinded in assigning the patients to the groups, they will not be blinded in the application and evaluation phase due to the application of virtual reality glasses. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported. Thus, the data analysis and statistics phase will also be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule. Patients in the study group will be shown a video with virtual reality glasses during the procedure. Patients will be asked to wear a virtual reality goggle (VR Box Virtual Reality Headset 3D Vr Glasses V2.0 2020 model) that is compatible with a mobile phone (Xiaomi Redmi Note 8 Pro 2019 model) with android operating system and minimizes sound loss in the supine position. With the virtual reality glasses, nature landscapes with relaxing music background will be watched by adjusting the volume at the level desired by the patient. Virtual reality glasses will be applied during the urodynamics procedure. After the device is applied to each patient, it will be disinfected in accordance with the company's recommendation.
  Interventions: Other: Virtual reality goggles
- CONTROL GROUP (No Intervention): The control group will receive routine care.

INTERVENTIONS:
Other: Virtual reality goggles — Patients in the study group will be shown a video with virtual reality glasses during the procedure. Patients will be asked to wear a virtual reality goggle (VR Box Virtual Reality Headset 3D Vr Glasses V2.0 2020 model) that is compatible with a mobile phone (Xiaomi Redmi Note 8 Pro 2019 model) with android operating system and minimizes sound loss in the supine position. With the virtual reality glasses, nature landscapes with relaxing music background will be watched by adjusting the volume at the level desired by the patient. Virtual reality goggles will be applied during the urodynamic procedure.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The research was planned as a randomized controlled experimental study to determine the effect of virtual reality goggles on pain, anxiety and hemodynamic variables during urodynamics. The minimum sample size was calculated as 42 in each group with d=0.8, (1- α, bidirectional), 95% power with reference to the effect size limit of 0.8 in G*Power (3.1) program. Descriptive Information Form, Visual Analog Scale, State Anxiety Scale and Hemodynamic Variables Monitoring Form will be used to collect research data. The individuals in the sample group will be informed about the method followed in the application and the research and their verbal and written permissions will be obtained. Introductory Information Form, Visual Analog Scale, State Anxiety Scale and Hemodynamic Variables Monitoring Form will be completed. After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule.Patients in the study group will be shown videos with virtual reality glasses during the procedure. Nature landscapes with relaxing music background will be watched with virtual reality goggles by adjusting the volume at the level desired by the patient. Virtual reality goggles will be applied during the urodynamic procedure. The control group will receive routine care. After the virtual reality application, pain, anxiety levels and hemodynamic variables will be re-evaluated immediately and 15 minutes after the procedure. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistical methods (number, percentage, min-max values, mean and standard deviation) will be used to evaluate the data. Parametric and nonparametric tests will be used according to the suitability of the data used for normal distribution. P < 0.05 will be taken as statistically significant difference

DETAILED DESCRIPTION:
The research was planned as a randomized controlled experimental study to determine the effect of virtual reality goggles on pain, anxiety and hemodynamic variables during urodynamics. The population of the study, which is planned as a randomized controlled experimental study, will consist of patients who apply to the Urology Outpatient Clinic of Mersin University Hospital and will undergo urodynamics. The minimum sample size was calculated as 42 in each group with d=0.8, (1- α, bidirectional), 95% power with reference to the effect size limit of 0.8 in G*Power (3.1) program. Descriptive Information Form, Visual Analog Scale, State Anxiety Scale and Hemodynamic Variables Monitoring Form will be used to collect research data. The individuals in the sample group will be informed about the method followed in the application and the research and their verbal and written permissions will be obtained. Introductory Information Form, Visual Analog Scale, State Anxiety Scale and Hemodynamic Variables Monitoring Form will be completed. After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule.Patients in the study group will be shown videos with virtual reality glasses during the procedure. Nature landscapes with relaxing music background will be watched with virtual reality goggles by adjusting the volume at the level desired by the patient. Virtual reality goggles will be applied during the urodynamic procedure. The control group will receive routine care. After the virtual reality application, pain, anxiety levels and hemodynamic variables will be re-evaluated immediately and 15 minutes after the procedure. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Pearson-χ2 test will be used for categorical variables. Descriptive statistical methods (number, percentage, min-max values, mean and standard deviation) will be used to evaluate the data. Parametric and nonparametric tests will be used according to the suitability of the data used for normal distribution. P < 0.05 will be taken as statistically significant difference

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study,
* between the ages of 18-65
* Conscious, oriented and cooperative,
* No communication problems,
* undergoing invasive urodynamics,
* No physical problems that would prevent the application of virtual reality goggles,
* No previous experience with virtual reality glasses,
* Undiagnosed anxiety,
* No medication for anxiety
* Patients without mental disorders

Exclusion Criteria:

* Who did not agree to participate in the study,
* Under 18 or over 65 years of age,
* Conscious, oriented and uncooperative,
* Communication problems,
* No invasive urodynamics procedure,
* Physical problem that would prevent the application of virtual reality goggles,
* Diagnosed with anxiety,
* Taking medication for anxiety (anxiolytics, antidepressants, antipsychotics, etc.),
* Patients with mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Pain score | 7 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no pain at all)-10 (very severe pain) to evaluate the level of pain (Wewers and Lowe, 1990).
Anxiety | 7 months
  The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Hemodynamic Variables | 7 months
  Hemodynamic Variables Monitoring Form : In this form, hemodynamic variables of the study and control groups measured before, immediately after and 15 minutes after the procedure will be recorded. Patient values will be measured and recorded by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, Principal Investigator — Mersin University; Elife KETTAŞ DÖLEK, Principal Investigator — Mersin Unıversity Hospital; Murat BOZLU, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biardeau X, Lam O, Ba V, Campeau L, Corcos J. Prospective evaluation of anxiety, pain, and embarrassment associated with cystoscopy and urodynamic testing in clinical practice. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):104-110. doi: 10.5489/cuaj.4127. PMID 28515809
- [Background] Dogan Yilmaz E, Unlusoy Dincer N. The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):318-328. doi: 10.1097/SGA.0000000000000733. Epub 2023 Jun 5. PMID 37278621
- [Background] Drake MJ, Doumouchtsis SK, Hashim H, Gammie A. Fundamentals of urodynamic practice, based on International Continence Society good urodynamic practices recommendations. Neurourol Urodyn. 2018 Aug;37(S6):S50-S60. doi: 10.1002/nau.23773. PMID 30614058
- [Background] Gammie A, Drake MJ. The fundamentals of uroflowmetry practice, based on International Continence Society good urodynamic practices recommendations. Neurourol Urodyn. 2018 Aug;37(S6):S44-S49. doi: 10.1002/nau.23777. PMID 30614059
- [Background] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973